CLINICAL TRIAL: NCT04052035
Title: Follicular Size and Ploidy: an Observational Study
Brief Title: Follicular Size and Ploidy Observational Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Daniela Nogueira, Consultant IVF Laboratory, ART Fertility Clinics LLC
Other Study IDs: 1905-ABU-061-ND
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Follicle Size; Age, Parental
Keywords: follicle size; maturity; euploid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — trophectoderm cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: measuring the size of the follicle at time of follicle aspiration — While for an OPU out of the study the follicles are aspirated without measuring their sizes, now the follicles will be measured before they are aspirated. The measurement of the follicles is a non- invasive measurement: as the OPU is always performed under vaginal echo-guidance, the follicles are visible on the screen connected to the vaginal echo probe. By measuring two dimensions of the follicle, an average follicle diameter is registered for that follicle

SUMMARY:
The primary objective is to determine which follicle sizes generate the highest rate of euploid blastocysts.

DETAILED DESCRIPTION:
The primary objective is to determine which follicle sizes generate the highest rate of euploid blastocysts.

Secondary objectives to be analysed between the different follicle sizes:

* The number of cumulus oocyte complexes (COCs) retrieved per aspirated follicle size
* The number of mature oocytes per COC retrieved (maturation rate)
* The number of normally fertilized oocytes per number of oocytes injected (fertilization rate)
* Embryo development up to the blastocyst stage
* Chromosomal status of the biopsied blastocysts
* Pregnancy rates after euploid blastocyst transfer
* Miscarriage rate after euploid blastocyst transfer

Most of the studies that looked at the relation between the follicular size and the developmental competence of the corresponding oocyte analysed normal responders with an average age of 35 years and normal BMI levels. However, during the last decades, a clear shift appeared in the patient population that present themselves for a fertility treatment. With many women delaying childbirth, we do not yet know how these advanced maternal age women may benefit from early or late trigger or from different follicular sizes.

Also, the rising prevalence of obesity may impact the follicular growth, which has not been analysed at the individual follicle size before.

For the above described reasons, we believe that the analysis of individual follicles and the developmental competence of the obtained oocyte, may guide us to improve individualized stimulation protocols for different subtypes of infertile patients. To guide us in this individualized process, this initial pilot study will be performed in a population of normal responders and will later be expanded to an infertile population with different characteristics.

ELIGIBILITY:
Inclusion Criteria:

Cycles with PGT-A analysis

* ICSI (intracytoplasmic sperm injection) only
* ICSI 40 hours after trigger
* Fresh oocytes
* Ejaculates: fresh or frozen: normozoospermia
* BMI ≤ 35kg/m 2
* Age ≤ 40 years
* AMH ≥ 1.1 ng/ml
* the number of follicles at the day of trigger: max 20 ≥ 11mm
* Stimulation protocol: Antagonist protocol with Menopur and and Dual trigger of (5.000-10.000IU) hCG and (0.2-0.3 mg) Gonapeptyl
* Final oocyte maturation trigger when 2-3 follicles reach size 17mm
* All races
* Embryo development in the Embryoscope with Global Total media

Exclusion Criteria:

* Inability to puncture all follicles from one ovary
* Endometriosis
* Hydrosalpinx
* History of uterine surgery
* History of previous treatment which may impact the ovarian reserve (adnexal surgery,
* chemotherapy, radiation…)
* Time between trigger and pick up deviating from 36 hours
* < 100.000 motile sperm
* Last follicular measurement day deviates more than 24 hours from the trigger day

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — it depends on the ability to produce follicles
Study Population: The study is eligible to all patients undergoing a fertility treatment with PGT-A analysis at the blastocyst stage
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Blastocyst ploidy outcome according to the follicular size at the OPU | 2 months
  Blastocyst ploidy is determined after biopsy of trophectoderm cells, taken from the blastocyst on day 5, 6 or 7 from development. A biopsy is only possible if an oocyte was retrieved from the follicle that was mature, normally fertilized and developed into a blastocyst of sufficient quality for biopsy).
  The following outcomes are possible:
  1. Normal
  2. Abnormal
  3. Inconclusive/No result

SECONDARY OUTCOMES:
Recovery rate | 2 months
  Number of COCs retrieved/ number of follicles aspirated
Maturate rate | 2 months
  # of MII oocytes/ # of COCs retrieved
Fertilization potential ( normal and abnormal fertilization) | 2 months
  Normal fertilization is assessed by the presence of 2 pronuclei 16-20 hours post insemination. This is normal fertilization. Abnormal fertilization is a deviation from the presence of 2 pronuclei, this can be one or three or more.
Embryo development up to blastocyst stage | 2 months
  development of an embryo from day 0 to the blastocyst stage includes all developmental stages The embryo will make multiple divisions that will be recorded every day of development. It wll go from 1 cell, to 2 cells, 3 cells etc to be 8 cells on day 3 of development. On day 4, the morula will form and the embryo will start to compact, which is indicated as compacting or compacted. After this stage, we are around day 5 of development, the embryo will start to cavitate, this is the beginning of blastulation. Different stages are observed. Bl1: cavity is less than 50%, bl2: cavity is larger tan 50%, bl3: full blastocyst, bl4; expanded blastocyst, bl5: hatching balstocyst, bl6: hatched blastocyst, bl7: hatching through an artificail opening, bl8: collpased blastocyst. Blastocysts will be scored according to Gardner and Schoolcraft (1999).
Embryo development in time lapse incubators | 2 months
  assessing all specific time points
Chromosomal status of biopsied embryos | 2 months
  Blastocysts of sufficient quality will undergo trophectoderm biopsy. These 4-8 cells that are taken from the embryo are genitically tested for their chromosomal copy number. This will give an indication on the genetic status of the embryo. The embryo will be euploid if 23 pairs of intact chromosomes are present. If not, they are aneuploid.
mtDNA copy number | 2 months
  Mitoscore values is the ratio of the mitochondrial DNA over the nuclear DNA. This is presented as a value and has been linked to the implantation potential of the embryo. There is no unit.
Miscarriage rate after single euploid embryo transfer | 2 months
  loss of a pregnancy with hcg levels above 1000 IU after transfer
pregnancy rate after euploid embryo transfer | 2 months
  presence of bhCG above 15IU 12 days after transfer
biochemical pregnancy rate | 2 months
  characterized only by the presence of bhCG above 15 IU, no presence of gestational sac
clinical pregnancy rate | 2 months
  hCG > 15 Iu/ml and ultrasound confirmation of a gestational sac
implantation rate | 2 months
  • Implantation rate calculated by the number of gestational sacs observed at echographic screening at 6 weeks of pregnancy divided by the number of embryos transferred, multiplied by 100.
ectopic pregnancy rate | 2 months
  where the embryo attached outside the uterus

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Elkhatib, MSc, Study Chair — IVIRMA Middle East Fertility Clinic
Locations (1):
- IVI Middle East Fertilty Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Information regarding the size of follicle and the PGT-A results will be shared through the discussion part.
  Further information regarding endocrine profile, fertilization and embryo development will be mentioned in the discussion as well, however, this data might be shared upon request after publication.
  Personal information such as Name and contact details will not be mentioned or shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Undecided
Access Criteria: Undecided